CLINICAL TRIAL: NCT01860001
Title: Incidence of Postoperative Ketosis and Metabolic Acidosis
Acronym: POKACID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR3828
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Metabolic Acidosis
Keywords: cancer; metabolic acidosis
MeSH Terms: conditions — Acidosis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to define the incidence and nature of acidosis after major surgery using Figge's equations to directly measure acidosis. This study will also aim to compare the ability of indirect measures (base deficit, anion gap,corrected anion gap and lactate) to identify the presence of tissue acids in this population. The incidence of postoperative ketoacidosis as a contributor to tissue acidosis will be assessed through the use of point of care urinalysis.

DETAILED DESCRIPTION:
Metabolic acidosis is a frequent occurrence following major surgery. Monitoring acid base disturbances and in particular diagnosing the aetiology of the acidosis are important parts of assessing a patient's cardiovascular status following surgery. The presence of a metabolic acidosis is frequently attributed to anaerobic metabolism leading to the generation of lactic acid due to hypovolaemia and poor tissue perfusion. This commonly results in clinicians treating postoperative patients with a metabolic acidosis by administering intravenous fluids containing 0.9% saline or Hartmann's solution (compound sodium lactate). If the cause of the metabolic acidosis is not hypovolaemia, treatment with intravenous fluids may actually exacerbate the acidosis by causing hyperchloraemia. An often overlooked cause of metabolic acidosis after surgery is starvation leading to ketoacidosis. All patients are starved for a minimum of six hours prior to general anaesthesia due to the potential risk of aspiration of gastric contents into the bronchial tree. Many patients are in fact fasted for much longer periods than this. There is, however, little data describing the incidence of ketoacidosis following surgery. In addition, there may be other causes of acidosis after surgery which often overlooked but can be determined using equations and mathematical models. The aim of this study is to define the incidence and nature of acidosis after major cancer surgery using using equations to directly determine acids. This study will also aim to compare the ability of commonly used indirect measures (base deficit, anion gap, corrected anion gap and lactate) to identify the presence of tissue acids in this population. The incidence of postoperative ketoacidosis as a contributor to tissue acidosis will be assessed through the use of point of care urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone major cancer surgery
* Patients who have an arterial line in place
* Patients who have a urinary catheter in place
* Patients who will be admitted to intensive care following surgery
* Adults >18 years
* Adults who are capable of reading and understanding English

Exclusion Criteria:

* Patient refusal
* Patients without an arterial line or urinary catheter in place
* Patients receiving glucose / sliding scale insulin for management of diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital patients seen in pre-operative assessment clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of tissue acidosis, defined as tissue acids > 5mEq/L (Figge's equation) within one hour of completion of surgery | 31/08/13

SECONDARY OUTCOMES:
Incidence of metabolic acidosis, defined by base deficit . 2 mEq/L (Henderson-Hasselback) within one hour of completion of surgery. | 31/08/13

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wigmore, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, England, United Kingdom